CLINICAL TRIAL: NCT06468540
Title: Comparative Study on the Efficacy of the Combination of Micropulse Laser With or Without Photodynamic Therapy in the Treatment of Chronic Central Serous Chorioretinal Disease
Brief Title: Combination of Micropulse Laser With or Without Photodynamic Therapy for Chronic Central Serous Chorioretinopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IIT-2024-04-376
Record Dates: First submitted 2024-06-08; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Central Serous Chorioretinopathy; Micropulse Laser; Photodynamic Therapy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, patients with chronic central serous chorioretinopathy who were treated by micropulse laser alone or micropulse laser combined with photodynamic therapy without drugs are retrospectively included. The visual acuity changes, subretinal fluid absorption and choroidal characteristics of the two groups are compared 1 to 6 months after treatment. We will also analyze baseline characteristics that influence post-treatment outcomes to identify potential predictors of poor treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* The patient diagnosed with chronic central serous chorioretinopathy with a history of more than 6 months. The diagnostic criteria for chronic CSC were as follows: FFA examination showed leakage of strong fluorescent spots with the extension of angiography time, and late fluorescence accumulation, accompanied by decreased central vision, darkening of vision, and deformable microopia. Fundus examination showed superficial detachment of retinal neuroepithelium in macula.
* Patients received single micropulse laser therapy or micropulse laser combined with drug-free photodynamic therapy, and had not received other laser or surgical treatment in the six months prior to treatment.
* Patients had follow-up data before and after treatment for 1 month and at least 6 months.

Exclusion Criteria:

* Patients with other fundus diseases or refractive interstitial opacity.
* During treatment, other treatments other than micropulse laser or drug-free photodynamic therapy were received.
* Various reasons led to incomplete patient data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient diagnosed with chronic central serous chorioretinopathy with a history of more than 6 months, who received single micropulse laser therapy or micropulse laser combined with drug-free photodynamic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
BCVA | 1 month and 6 months
  Best-corrected visual acuity using logMAR
CRT | 1 month and 6 months
  Central retinal thickness on OCT

SECONDARY OUTCOMES:
SFCT | 1 month and 6 months
  subfoveal choroidal thickness on OCTA